CLINICAL TRIAL: NCT02275429
Title: Etude Des Troubles métaboliques Induits Par Une Course à Pied très Longue Distance, " La Diagonale Des Fous " de La Réunion / Metabolic Disorders in Ultramarathon Runners of the Madmen's Diagonal Race on Reunion Island
Brief Title: Metabolic Disorders in Ultramarathon Runners During and After the Reunion Island Madmen's Diagonal
Acronym: METARUN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de la Réunion (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014/CHU/03
Record Dates: First submitted 2014-10-15; First posted 2014-10-27 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Metabolic Diseases
Keywords: Metabolic Diseases; Athletes; Running; Selenium; Zinc; Iron Metabolism Disorders; Water-Electrolyte Imbalance; Hyperkalemia; Hypernatremia; Selenium levels before and after the race; Levels of other electrolytes and markers
MeSH Terms: conditions — Metabolic Diseases; Iron Metabolism Disorders; Water-Electrolyte Imbalance; Hyperkalemia; Hypernatremia | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Runners (Other): Each year, about 1,200 runners residing on Reunion Island take the start of the Madmen's Diagonal ultramarathon. Among those, 500 runners will be selected at random and will receive a letter informing them of the study and requesting their participation. Those who accept are to contact the study team. Among those volunteers, 100 runners will be selected randomly and included in the study. They will undergo a blood test the day before the race starts (day 0, when they retrieve their race number), upon completion of the race, and upon days 7 and 28.
  Interventions: Procedure: Blood test

INTERVENTIONS:
Procedure: Blood test — blood will be drawn the day before the race (day 0), upon completion of the race (between 27 and 67 hours after departure), and on days 7 and 28

SUMMARY:
Acute consequences of ultramarathon running are still unknown as very little research has been done on the matter. The investigators will assess the consequences on the metabolism of runners in the ultramarathon Madmen's Diagonal on Reunion Island. Data from the literature suggest that runners undergo loss of zinc, copper, iron, magnesium not unlike the loss of metabolites in systemic inflammatory response syndrome. The purpose of this study is to assess the metabolic disorders (selenium, zinc, vitamins B9 and B12) in ultramarathon runners, during and up to 28 days after the Madmen's Diagonal which takes place on Reunion Island every year in October.

DETAILED DESCRIPTION:
Ultramarathons are races involving walking or running longer than the traditional marathon length of 42km and frequently take longer than 12 hours to complete. These races are increasingly frequent and racers attempt to push back the limits of what their body can accomplish. However, these races are not without certain risks.

The Reunion Island Grand Raid (or Madmen's Diagonal) is one such race, crossing the island over 163 km (101 mi) with an altitude gain of 9,643 meters (31,637 ft). Temperatures vary from 0 et 30 degrees Celsius (32-86°F) and the race can take 27 to 67 hours to complete. About 40% of the racers do not cross the finish line. Each year, two or three racers are hospitalized each year in the intensive care unit (ICU) for tubular necrosis and treated with dialysis. Scientific literature shows that racers can present acute rhabdomyolysis, with elevated levels of CPK-MB. Nevertheless, there have been very few studies on the impact of these ultramarathon racers on other biological parameters. As the racers compete and lose about a liter of sweat every hour, they also lose ions and trace metals such as zinc, copper, iron, magnesium, which can have major repercussions during and after the race. These losses are akin to those observed in severe burn victims. In these patients, it has been shown that supplementation in trace elements can decrease mortality and hospitalization time.

Moreover, a major inflammatory response has been observed in racers who compete in ultramarathons. This inflammatory response is similar to that of the systemic inflammatory response syndrome (SIRS). Patients in the ICU who are septic or who present a SIRS also have metabolic diseases, and it has been shown that selenium levels are a prognostic factor of SIRS and supplementation can increase survival rates.

Investigators present the hypothesis that ultramarathon racers can have decreased levels of selenium and other ions and trace metals and that specific supplementation can limit risks and improve recovery. More specifically, investigators suggest that selenium levels will decrease by 25% after the race and remain so at least a week.

ELIGIBILITY:
Inclusion Criteria:

* Ultramarathon runner in the Madmen's Diagonal on Reunion Island (October 2014 )
* Aged 18 years or older
* Lives on Reunion Island
* Gave informed consent
* Medical certificate allowing the participation in an ultramarathon

Exclusion Criteria:

* Aged less than 18 years Ultramarathon runner in the Bourbon Trail or Mascarenes races (which take place at the same time as the Madmen's Diagonal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2014-10; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Assess the selenium levels | 28 days
  Blood wil be analyzed prior to the start of the race, upon completion of the race (anywhere between 27 and 67 hours after the start of the race), and upon days 7 and 28. Blood will be drawn in the same medical laboratory at the Reunion Island University Hospital site of Saint Denis.

SECONDARY OUTCOMES:
- Assess Ions and trace metals (Sodium, Potassium, Chloride, Zinc) | 28 days
- Assess Renal function tests (creatinine, blood urea nitrogen) | 28 days
- Assess liver function (total protein, cardiac markers (myoglobin, CPK-MB) | 28 days
- Assess iron and ferritin | 28 days
- Assess blood disorder (vitamin B12, folic acid or vitamin B9) | 28 days
- Assess hematology disorder | 28 days
Fatigue assessment: assessed via a visual analogue scale | 28 days
  Fatigue will be assessed via a visual analogue scale

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme SUDRIAL, MD, Principal Investigator — CHU Réunion
Locations (1):
- Reunion Island University Hospital, Saint-Denis, Reunion Island, France